CLINICAL TRIAL: NCT03177967
Title: "Get up" - The Sleep Study in Oppegard (Stå Opp - Søvnstudien i Oppegård)
Brief Title: "Get up" - The Sleep Study in Oppegard
Acronym: Stå Opp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017/462
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; Cognitive behavioral treatment for insomnia (CBT-I)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment groups spring (1,2) (Experimental): Seven sessions CBT-I treatment for two different groups of eight participants (n=16)
  Interventions: Sleep restriction/Stimulus Control Discussion of adverse cognitions about sleep
  Interventions: Behavioral: Sleep Restriction Therapy/Stimulus Control; Other: Discussions about adverse cognitions about sleep
- Waiting list - Treatment groups fall (Experimental): This group (n=22) receives no treatment during the spring and summer, and is measured three times as a waiting list control in this period of time. The same group will receive treatment i three different groups during sept/oct.
  Interventions: Sleep restriction/Stimulus Control Discussion of adverse cognitions about sleep
  Interventions: Behavioral: Sleep Restriction Therapy/Stimulus Control; Other: Discussions about adverse cognitions about sleep
- Psychoeducative course in Nesodden (Active Comparator): This group (expected to be n=16) will receive a four session psychoeducative learning based course on how to manage insomnia
  Interventions: Psychoeducative advice to improve sleep
  Interventions: Other: Psychoeducative advice about how to improve sleep

INTERVENTIONS:
Behavioral: Sleep Restriction Therapy/Stimulus Control — Sleep Restriction Therapy focuses on forcing your available sleep time into a fixed window. The sleeper sets a bedtime and wake-up time and sticks to those times closely. The time allocated for being allowed in bed is determined from an estimate of how long the patient in average has been sleeping during the night, in the week before treatment. The goal is to have the patient sleeping the entire time he or she is in bed by making this period so restricted that the patient has no chance of sleeping enough. Once this goal is achieved, the time allocated for bed can be slowly increased, for example by 15 minutes at a time. After enough iterations, an equilibrium is achieved that the patient can keep maintaining after treatment has completed.
  Arms: Treatment groups spring (1,2); Waiting list - Treatment groups fall
Other: Discussions about adverse cognitions about sleep — Group discussions about insomnia, CBT-i treatment and it's effects
  Arms: Treatment groups spring (1,2); Waiting list - Treatment groups fall
Other: Psychoeducative advice about how to improve sleep — Learning about sleep and sleep hygiene tips. It also includes learning about stimulus control and sleep restriction.
  Arms: Psychoeducative course in Nesodden

SUMMARY:
A randomized, controlled study to examine the effect of group treatment for insomnia (CBT-I) in an outpatient clinic compared with waiting list and treatment-as-usual (sleep-hygiene based educational course)

DETAILED DESCRIPTION:
Insomnia is a large public health concern with latest reports pointing to almost 15 % of the population in Norway having insomnia (Pallesen, Sivertsen, Nordhus, & Bjorvatn, 2014). At the same time there is a scientific consensus about how to best treat insomnia (CBT-I), and it is empirically proven that this is quite effective treatment (Okajima, Komada & Inoue, 2011).

We therefore want to conduct a study to examine if CBT-I treatment in an public outpatient clinic is effective compared with waiting list and a psychoeducational course.

The design is a randomized controlled study with three different conditions (CBT-I versus waiting list versus TAU) that will be compared over time. We will use an A-B-design which can effectively compare the different conditions in the study. We have recruited a total of 62 patients, and completed a individual session with each of these individuals resulting in a total admission of 38 participants in the study. The remaining 24 patients either didn't fit the selection criteria, or we were unable to get in touch with them to agree on an appointment.

Of the 38 participants enrolled in the study, 16 will get CBT-I, Group based treatment during May and June of 2017 (a total of seven sessions over nine weeks), and the remaining 22 will get the same treatment in September and October 2017. The maximum number of patients per group is eight (8) and we randomized whether participants got assigned to treatment in May/June or September/October.

We measure all participants at the individual pre-screening (T1), Treatment Group 1 and 2 gets treatment in May and June and will be measured in every other treatment session (2,4,6 and 7) From now on called (T2, T3, T4, T5). Treatment Group 3,4 and 5 (all getting treatment i September/October) is measured at T2 and T5. T1 was conducted during the last week of April and T5 is towards the end of June 2017.

Treatment Group 3, 4 and 5 will start their treatment and be measured at session 2 (T6) in mid-September, and Treatment Group 1 and 2 will also be measured at this point. Treatment Group 3, 4 and 5 will then be measured at treatment session 4,6 and 7, just like treatment Group 1 and 2 was during their treatment. (From now on T7, T8, T9). Treatment Groups 1 and 2 will also be measured at T9.

The treatment-as-usual condition is conducted in Nesodden kommune, and it is a psychoeducative, learning based course. This course consists of 4 sessions, and the participants is measured at session 1,3 and 4 in addition to a 6 months follow-up measure. They also get measured at pre-screening. We expect about 16 participants to complete this course.

ELIGIBILITY:
Inclusion Criteria:

* persons above the age of 18
* living in the municipalities of Oppegård and Ski
* fits the criteria for moderate or severe clinical insomnia, as measured by Insomnia Severity Index (Bastien C. H., Valliéres A., Morin C. M., 2001)

Exclusion Criteria:

* bipolar disorder
* epilepsy
* severe depressive episode
* psychosis disorders
* somatic sleep disorders (untreated sleep apnea, restless leg syndrome, narcolepsy, and sleepwalking)
* persons with a high risk of falling at home
* persons handling heavy machinery
* severe personality disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | We expect the decline in insomnia symptoms to start by session four (late may, 2017), and continue through session six (medio june, 2017) and seven (late june, 2017), and to be maintained at six-months follow up (november, 2017).
  Reduction in score on the Insomnia Severity Index

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-item Scale (GAD-7) | We expect the decline in anxiety symptoms to start declining by session four (late may, 2017), and to be maintained at six-months follow up (november, 2017).
  Reduction in anxiety symptoms by the end of the treatment period
The Patient Health Questionnaire (PHQ-9) | We expect the decline in symptoms of depression to start declining by session four (late may, 2017), and to be maintained at six-months follow up (november, 2017).
  Reduction in symptoms of depression by the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Knut Inge Klepp, PhD, Study Chair — Executive director
Locations (1):
- Oppegård kommune, Kolbotn, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okajima, I., Komada, Y. and Inoue, Y. (2011), A meta-analysis on the treatment effectiveness of cognitive behavioral therapy for primary insomnia. Sleep and Biological Rhythms, 9: 24-34. doi:10.1111/j.1479-8425.2010.00481.x
- [Background] Pallesen S, Sivertsen B, Nordhus IH, Bjorvatn B. A 10-year trend of insomnia prevalence in the adult Norwegian population. Sleep Med. 2014 Feb;15(2):173-9. doi: 10.1016/j.sleep.2013.10.009. Epub 2013 Dec 1. PMID 24382513
- [Background] Kessler RC, Berglund PA, Coulouvrat C, Hajak G, Roth T, Shahly V, Shillington AC, Stephenson JJ, Walsh JK. Insomnia and the performance of US workers: results from the America insomnia survey. Sleep. 2011 Sep 1;34(9):1161-71. doi: 10.5665/SLEEP.1230. PMID 21886353
- [Background] Sivertsen B, Salo P, Mykletun A, Hysing M, Pallesen S, Krokstad S, Nordhus IH, Overland S. The bidirectional association between depression and insomnia: the HUNT study. Psychosom Med. 2012 Sep;74(7):758-65. doi: 10.1097/PSY.0b013e3182648619. Epub 2012 Aug 9. PMID 22879427
- [Background] Irwin MR, Cole JC, Nicassio PM. Comparative meta-analysis of behavioral interventions for insomnia and their efficacy in middle-aged adults and in older adults 55+ years of age. Health Psychol. 2006 Jan;25(1):3-14. doi: 10.1037/0278-6133.25.1.3. PMID 16448292
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Falloon K, Elley CR, Fernando A 3rd, Lee AC, Arroll B. Simplified sleep restriction for insomnia in general practice: a randomised controlled trial. Br J Gen Pract. 2015 Aug;65(637):e508-15. doi: 10.3399/bjgp15X686137. PMID 26212846